CLINICAL TRIAL: NCT04648111
Title: Implementing Peri-operative Mobile Application for Contactless Screening and Vital Signs Measurement (MAC-VITAL): A Proof of Concept Trial
Brief Title: Implementing Peri-operative Mobile Application for Contactless Vital Signs
Acronym: MAC-VITAL
Status: Completed | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Dr. Frances Chung, Anesthesiologist, University Health Network, Toronto
Other Study IDs: UHN CAPCR#20-5683
Record Dates: First submitted 2020-11-13; First posted 2020-12-01 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-11

CONDITIONS: Blood Pressure, Heart Rate, Breathing Rate and Oxygen Level
MeSH Terms: interventions — Vital Signs

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Vital sign measurement — Vital signs measurement will be obtained by the research staff using hospital standard medical devices and the Anura Research App will also be used to measure vital signs. Measurement will take place before surgery and post surgery (1 ±2hrs and 2 ±4hrs after surgery).

SUMMARY:
The huge impact of the COVID-19 pandemic on global healthcare systems has prompted search for novel tools to stem the tide. New digital health tools can provide possible health solutions in this time of unprecedented medical crisis to mitigate the impact of this pandemic. This proof of concept study will determine the feasibility and effectiveness of implementing a mobile application for contactless measurement of vital signs (MAC-VITAL) such as blood pressure (BP), heart rate (HR), respiratory rate (RR) and oxyhemoglobin saturation (SpO2) from surgical patients peri-operatively. Contactless measurement of vital signs will bridge the current gap between virtual care and in-person medical assessments. This study aims to determine whether a mobile app can effectively measure vital signs without any person to person contact and how this technology can be implemented in a peri-operative setting during COVID-19.

DETAILED DESCRIPTION:
This study is a prospective proof of concept study to be conducted at Toronto Western Hospital,Toronto General Hospital, Hamilton General Hospital (Hamilton, Ontario), Juravinski Hospital (Hamilton, Ontario) and Trillium Health Partners, Mississauga, Ontario. This proof of concept study will determine the feasibility and effectiveness of implementing a contactless mobile application to obtain vital signs from patients in the peri-operative setting. Informed consent to participate in the study will be obtained.

Vital signs measurement will be obtained by the research staff using hospital standard medical devices and the Anura Research App will also be used to measure vital signs. Measurement will take place before surgery and post surgery (1 ±2hrs and 2 ±4hrs after surgery).

ELIGIBILITY:
Inclusion Criteria

* Patients scheduled to undergoing elective inpatient surgery under general and/or regional anesthesia
* 18 years or older

Exclusion Criteria

* Refusal to consent for the study
* Non-English speaking.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled to undergoing elective inpatient surgery under general and/or regional anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 91 (Actual)
Dates: Start 2021-06-04 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Vital signs measurement | 24 hours
  Blood pressure will be measured by using both AnuraTM research app and standard medical grade Blood pressure machine pre-and post-operatively.
Vital signs measurement | 24 hours
  Heart rate will be measured by using both AnuraTM research app and standard medical grade Blood pressure machine pre-and post-operatively.
Vital signs measurement | 24 hours
  Breathing rate will be measured by using both AnuraTM research app and standard medical grade Blood pressure machine pre-and post-operatively.
Vital signs measurement | 24 hours
  Heart rate variability will be measured by using both AnuraTM research app and standard medical grade Blood pressure machine pre-and post-operatively.
Vital signs measurement | 24 hours
  Oxygen saturation will be measured by using both AnuraTM research app and standard medical grade Blood pressure machine pre-and post-operatively.

CONTACTS AND LOCATIONS:
Locations (1):
- 399 Bathurst St.,Toronto Western Hopsital, Preadmission Clinic, Dept. of Anesthesia, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No